CLINICAL TRIAL: NCT07087847
Title: Prospective, Single-Center, Single-Arm Clinical Study of Ex Vivo T-Cell-Depleted Haploidentical Transplantation Bridging With Chimeric Antigen Receptor T-cell Therapy and Prophylactic Memory T Cell Infusion for Acute Leukemia
Brief Title: Ex Vivo T-Cell-Depleted Haploidentical Transplantation Bridging With Chimeric Antigen Receptor T-cell Therapy and Prophylactic Memory T Cell Infusion for Acute Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Miltenyi Biotec B.V. & Co. KG (Industry)
Responsible Party: Principal Investigator, Hu Xiaoxia, Professor of hematology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-TCD-2025
Record Dates: First submitted 2025-07-15; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Acute Leukemia; Acute Leukemia Refractory; Acute Myeloid Leukemia (AML); ALL (Acute B-Lymphoblastic Leukemia); Acute Leukemia in Relapse
Keywords: ex vivo t cell depletion; TCRab depletion; CD45RA depletion; memory T cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: open, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCRαβ+/CD45RA+ depleted haplo-HSCT bridging with CAR-T (Experimental): For patients with refractory/relapsed (R/R) leukemia:
  Approximately 28 days post-CAR-T therapy, a hematologic assessment will be performed. Eligible patients meeting the inclusion criteria will subsequently undergo TCRαβ+/CD45RA+-depleted haploidentical hematopoietic stem cell transplantation (haplo-HSCT).
  Interventions: Biological: TCRαβ+/CD45RA+depleted haploidentical hematopoietic stem cell transplantation (haplo-HSCT)

INTERVENTIONS:
Biological: TCRαβ+/CD45RA+depleted haploidentical hematopoietic stem cell transplantation (haplo-HSCT) — Approximately 28 days post-CAR-T therapy, a hematologic assessment will be performed. Eligible patients meeting the inclusion criteria will subsequently undergo TCRαβ+/CD45RA+depleted haploidentical hematopoietic stem cell transplantation (haplo-HSCT).Collect peripheral blood stem cells (PBSC) from the haplo-donor.Split the graft into two fractions at a 9:1 ratio, 90% fraction: subject to TCRαβ+ T-cell depletion, 10% fraction: subject to CD45RA+ T-cell depletion. Primary graft (TCRαβ+depleted and partial CD45RA+ depleted): Freshly infused into the recipient. Residual CD45RA-depleted lymphocytes: Cryopreserved for prophylactic donor lymphocyte infusion (DLI) as needed.

SUMMARY:
CAR-T therapy has evolved as a pivotal treatment for relapsed/refractory (R/R) leukemia, demonstrating improved remission rates and manageable adverse events. However, over 50% of patients achieving complete remission (CR) experience relapse within one year (1-year cumulative incidence rate, CIR) due to antigen escape, CAR-T functional exhaustion, premature cell depletion, and immunosuppressive microenvironments. Novel strategies are urgently needed to sustain durable responses.

Bridging CAR-T therapy with TCRαβ+ and CD45RA+ cell-depleted haploidentical hematopoietic stem cell transplantation (HSCT) offers dual benefits: Graft-versus-leukemia (GvL) effects mediated by donor-derived NK cells and γδT cells target non-CAR-dependent antigens, mitigating immune evasion. Rapid hematopoietic reconstitution reduces prolonged cytopenia-related complications from prior therapies. This protocol further incorporates prophylactic CD45RO+ memory T-cell (Tm) infusion to: Minimize graft-versus-host disease (GVHD) risks compared to conventional donor lymphocyte infusion (DLI). Enhance adoptive immunity against infections/relapse via transferred donor memory immunity. We design this prospective, single-center, single-arm trial to evaluate the efficacy/safety of this approach using the CliniMACS® system for ex vivo TCRαβ+/CD45RA+ depletion in R/R leukemia patients post-CAR-T.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients with refractory or relapsed (R/R) leukemia.
* Donor Availability: No matched sibling or unrelated donor identified through HLA typing.
* Disease Status Post-CAR-T: including achieved complete remission (CR), minimal residual disease (MRD)-negative in bone marrow and no extramedullary relapse.
* Normal Organ Function (meeting the following criteria): including liver function: ALT/AST ≤10×ULN (upper limit of normal), total bilirubin (TBIL) ≤5×ULN, renal function: BUN and serum creatinine (Cr) ≤1.25×ULN and cardiac function: No evidence of cardiac insufficiency (confirmed by ECG and echocardiography).
* Informed Consent: a signed informed consent form (ICF) is obtained

Exclusion Criteria:

* Presence of any absolute contraindication to hematopoietic stem cell transplantation.
* Severe Comorbidities with Major Organ Dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
2-Year Event-Free Survival (EFS) Rate | 2 years
  Definition: The proportion of patients who remain free from any of the following events for 2 years post-transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No